CLINICAL TRIAL: NCT05452070
Title: An International, Multicenter, Evaluator-blinded, Randomized, Parallel-Group, Controlled Study of the Safety and Effectiveness of HArmonyCa Lidocaine Injectable Gel for Mid Face Soft Tissue Augmentation
Brief Title: A Study to Assess Adverse Events and Change in Disease Activity of HArmonyCa Lidocaine Injectable Gel for Mid Face Soft Tissue Augmentation in Adult Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M21-784
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Mid Face Volume Deficit

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HArmonyCa Lidocaine Injectable Gel (Experimental): Participants will receive HArmonyCa Lidocaine Injectable Gel on Day 1 and followed for up to 25 months. Participants will have the opportunity to receive optional touch-up and optional repeat treatment of HArmonyCa Lidocaine injectable gel during the follow-up duration period.
  Interventions: Device: HArmonyCa Lidocaine Injectable Gel
- Control Group (Other): Participants will be followed for 3 months. Participants can opt to receive HArmonyCa Lidocaine Injectable Gel after 3 months and followed for up to 25 months.
  Interventions: Device: HArmonyCa Lidocaine Injectable Gel

INTERVENTIONS:
Device: HArmonyCa Lidocaine Injectable Gel — Subdermal or deep dermal injection

SUMMARY:
The cumulative effect of aging and environmental exposures (ie, ultraviolet, infrared, and visible light radiation and pollution) leads to wrinkles, discoloration, laxity, and roughness of sun exposed skin. The rapid restoration of soft tissue augmentation is commonly achieved by the use of dermal fillers. HArmonyCa Lidocaine injectable gel is a dermal filler intended for facial soft tissue augmentation. The purpose of this study is to assess adverse events and effectiveness of HArmonyCa Lidocaine injectable gel in adults seeking mid face soft tissue augmentation.

HArmonyCa Lidocaine Injectable Gel is an investigational device being developed for soft tissue augmentation in the mid face. Participants are placed in 1 of 2 groups, called treatment arms. There is a 1 in 3 chance that participants will be assigned to the control group. Around 160 adult participants seeking soft tissue augmentation will be enrolled in the study at approximately 15 sites worldwide.

Participants in the treatment group will receive HArmonyCa Lidocaine injectable gel at Day 1 and followed for up to 25 Months. Participants will have the opportunity to receive optional touch-up and optional repeat treatment of HArmonyCa Lidocaine injectable gel during the follow-up duration period. Participants in the control group are followed for 3 months and then can opt to receive HArmonyCa Lidocaine Injectable Gel at the end of month 3. The control group will participate in the study for up to 25 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be in general good health.
* Participant seeking soft tissue augmentation in the mid face.
* Participant must be capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in the protocol.
* Able, as assessed by the TI, and willing to follow study instructions (including compliance with the safety e-diary) and likely to complete all required study visits.

Exclusion Criteria:

* Has experienced trauma to the face within 6 months before enrollment or has residual deficiencies, deformities, or scarring
* Has active or recurrent inflammation or infection in either eye
* Has tendency to develop hypertrophic scarring and/or keloid scarring
* Has active autoimmune disease
* Has current cutaneous or mucosal inflammatory or infectious processes (eg, acne, herpes), abscess, an unhealed wound, or a cancerous or precancerous lesion, in the face
* Has fat injection or permanent facial implants (eg, polymethylmethacrylate, silicone, polytetrafluoroethylene) anywhere in the face
* Has temporary dermal filler injections in the face within 24 months before enrollment
* Has semi-permanent fillers (eg, poly-L-lactic acid, CaHA) anywhere in the face within 36 months before enrollment
* Has botulinum toxin treatment in cheek area (including crow's feet) within 6 months before enrollment
* Has mesotherapy or cosmetic facial procedures in the face within 6 months before enrollment. Examples of mesotherapy or cosmetic facial procedures are face-lift, laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, moderate or greater depth chemical peel, or other ablative procedures
* Has tattoos, piercings, facial hair, (unless willing to remove prior to each assessment visit) or scars in the face that would interfere with the visualization of the face for the effectiveness assessment
* Undergone a dental procedure within 6 weeks before treatment or plan to undergo a dental procedure (other than prophylaxis or dental fillings) during the course of the study
* History of an allergic reaction or significant sensitivity to constituents of the study investigational product (and its excipients) and/or other products in the same class (lidocaine [or any amide-based anesthetics], HA products, or Streptococcal protein).
* Any investigational treatment within 30 days or 5 half-lives of the treatment (whichever is longer) prior to the first dose of study treatment or is currently enrolled in another clinical study.
* Any live vaccine within 4 weeks prior to the first dose of study treatment, or expected need of live vaccination during study participation including at least 4 weeks after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving "Responder" Status for Evaluating Investigator's (EI) live assessment of Mid Face Volume Deficit Scale (MFVDS) | Month 3
  A "responder" is a participant with at least 1- grade improvement (reduction) of mid face soft tissue deficit using the MFVDS. MFVDS is a validated 6-point scale (0 = None, 5 = Severe).
Number of Participants with Adverse Events | Up to 25 Months
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug.

SECONDARY OUTCOMES:
Percentage of Participants Achieving "Responder" Status for EI's Live Assessment of Global Aesthetic Improvement Scale (GAIS). | Month 3
  A "responder" is a participant who achieves improved or much improved on GAIS. GAIS is a 5-point scale used to assess global aesthetic improvement of the cheek area (2=Much Improved, -2=Much Worse).
Percentage of Participants Achieving "Responder" Status for Participant Assessment of Global Aesthetic Improvement Scale (GAIS). | Month 3
  A "responder" is a participant who achieves improved or much improved on GAIS. GAIS is a 5-point scale used to assess global aesthetic improvement of the cheek area (2=Much Improved, -2=Much Worse).
Change from baseline on overall score in FACE-Q Satisfaction with cheeks specific questionnaire | Month 3
  In the FACE-Q Satisfaction with Cheeks questionnaire, the responses will be summed and converted to a Rasch-transformed score that ranges from 0 to 100.
Change from baseline on overall score in FACE-Q Satisfaction with lower face and jawline specific questionnaire | Month 3
  In the FACE-Q Satisfaction with lower face and jawline specific questionnaire, the responses will be summed and converted to a Rasch-transformed score that ranges from 0 to 100.
Change from baseline on overall score in FACE-Q Satisfaction with appearance specific questionnaire | Month 3
  In the FACE-Q Satisfaction with appearance specific questionnaire, the responses will be summed and converted to a Rasch-transformed score that ranges from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (12):
- Canada (8):
  - YVR Aesthetics Training & Study Centre /ID# 239809, Vancouver, British Columbia
  - Humphrey & Beleznay Cosmetic Dermatology /ID# 239805, Vancouver, British Columbia
  - Pacific Derm /ID# 240785, Vancouver, British Columbia
  - Skin Matters Medical Aesthetic Centre /ID# 239986, Vancouver, British Columbia
  - Dermetics Cosmetic Dermatology /ID# 246536, Burlington, Ontario
  - The Centre for Clinical Trials /ID# 246409, Oakville, Ontario
  - Bertucci MedSpa Inc. /ID# 246496, Woodbridge, Ontario
  - Erevna Innovations Inc. /ID# 240401, Westmount, Quebec
- Spain (2):
  - Instituto Medico Miramar /ID# 240939, Málaga, Malaga
  - WM Hospitals /ID# 245747, Barcelona
- United Kingdom (2):
  - Dr Nestor's Medical Cosmetic Centre /ID# 246406, Edinburgh
  - MediZen /ID# 240102, Sutton Coldfield

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/